CLINICAL TRIAL: NCT04847310
Title: Cost-effectiveness and Cost-Utility Evaluation of the Individual vs. Group Transdiagnostic Psychological Treatment for Emotional Disorders in Primary Care (PsicAP-Costs)
Brief Title: Cost-benefit Evaluation of a Transdiagnostic Psychological Treatment for Emotional Disorders in Primary Care
Acronym: PsicAP-Costs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: State Research Agency, Spain (Other Government)
Responsible Party: Principal Investigator, Ángel Aguilera Martín, Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2019-107243RB-C22
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Emotional Disorder; Depression; Somatoform Disorders; Anxiety Disorders
Keywords: transdiagnostic therapy; emotional disorders; primary care; cost-benefit analysis; brief psychological treatments; randomized controlled trial; depression; anxiety disorders; somatoform disorders
MeSH Terms: conditions — Depression; Somatoform Disorders; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial with pre-post measures and follow-ups.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded during pre- and post-treatment. Participants will be blinded during pretreatment assessment; however, it cannot be guaranteed that they will keep blinded in post-treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Other: Group brief transdiagnostic cognitive-behavioral therapy
- Group 2 (Experimental)
  Interventions: Other: Individual brief transdiagnostic cognitive-behavioral therapy
- Group 3 (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Group brief transdiagnostic cognitive-behavioral therapy — An adaptation of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) (Barlow et al., 2015) and the IAPT programme (Clark, 2018). It has been developed by Cano-Vindel (González-Blanch et al., 2018) and consists in seven 90-minute sessions, provided by a non-assessor clinical psychologist in 12-16 weeks, with 8-10 participants per group. Sessions are weekly or biweekly, reducing their frequency as the intervention advances. The activities and homework proposed are supported with materials such as theory documents, a CD for progressive muscle relaxation, self-recording sheets, and a therapy web (www.desordenesemocionales.es).
  Other Names: Group tCBT
  Arms: Group 1
Other: Individual brief transdiagnostic cognitive-behavioral therapy — An adaption of the group therapy, with the same phases. However, since it is an individual intervention, it is more flexible than group one and its contents and duration can be personalized. This intervention consists of a minimum of 6 and a maximum of 8 sessions of 30-60 minutes, provided by a clinical psychologist not involved in the assessments.
  Other Names: Individual tCBT
  Arms: Group 2
Other: Treatment as usual — Participants in this group will be provided the common primary care treatment by the GP, in a face-to-face consultation that seldom exceeds 10 minutes. TAU usually consists in pharmacological treatment prescribed by the GP, however, it might also consist in practical advice or even non-treatment (Watts et al., 2015). The first consultation will count as part of the recruitment process and, if the patient accepts to participate in the trial, no therapeutic help will be provided to them until they are allocated. Once in the TAU intervention, if the practitioner recommended any psychological treatment as part of it (e.g., referral to specialized care), the participant would be excluded to avoid contamination between clusters. TAU has not a specific amount of sessions; it will finish when the GP considers the patient is recovered.
  Other Names: TAU
  Arms: Group 3

SUMMARY:
The aim of this study is to compare, in cost-effectiveness and cost-utility terms, a brief transdiagnostic cognitive-behavioural therapy in two different modes, individual and group, with the treatment usually administered in primary care (TAU).

Participants between 18 and 65 years old and with, according to the pretreatment evaluation, mild to moderate emotional disorders will be randomly allocated to the three clusters. They will be assessed again immediately after treatment and 6 and 12 months later.

The study hypotheses expect to find (H1) the individual treatment generally as effective as the group one, whereas (H2) the TAU will be the least effective. (H3) The group therapy is expected to get the best results in terms of cost-effectiveness and (H4) the TAU will get the worst cost-effectiveness results. Furthermore, (H5) it is expected to find these results across the follow-up assessments too.

ELIGIBILITY:
Inclusion Criteria:

* Mild/moderate emotional disorder

Exclusion Criteria:

* Severe mental disorder (including severe depressive or anxiety disorders, not somatizations)
* High level of impairment
* Recent, severe suicide attempt
* No emotional disorder/Below the instruments cut-off points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms: 9-item Patient Health Questionnaire (PHQ-9) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The PHQ-9 (Kroenke et al., 2001) is the depression module of the PHQ (Díez-Quevedo et al., 2001; Spitzer et al., 1999), that scores the 9 DSM-IV depression criteria present in the last two weeks from 0 ("not at all") to 3 ("nearly every day"). A score of 10 is usually set as the cut-off point for major depression disorder (MDD): a score of 10-14 indicates minor depression, moderate MDD, or dysthymia; 15-19, moderately severe MDD; and 20-27, severe MDD. This tool has been tested in Spanish primary care centres (McDonald's ω = .89) (Muñoz-Navarro, Cano-Vindel, Medrano et al., 2017), finding 12 as the best cut point for MDD diagnosis (sensitivity of 84% and specificity of 78%) compared with 10 (sensitivity of 95% and specificity of 67%).
Change in anxiety symptoms: 7-item General Anxiety Disorder scale (GAD-7) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The GAD-7 (Spitzer et al., 2006) assesses common anxiety symptoms in the last two weeks, scoring from 0 ("not at all") to 3 ("nearly every day"). Cut points of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively. The algorithm sets 8 as the cut point for GAD, however it has been found that a score of 10 is more optimal (Spitzer et al., 2006). We will use the version validated by García-Campayo et al. (2010), that was recently tested in primary care centres (Cronbach's α = .83) (Muñoz-Navarro, Cano-Vindel, Moriana et al., 2017), confirming the score of 10 as the best diagnostic criterion (sensitivity of 87% and specificity of 78%).
Change in panic symptoms: Patient Health Questionnaire-Panic Disorder (PHQ-PD) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The PHQ-PD is the specific panic disorder module of the PHQ and scores each DSM-IV criterion as "yes" or "no" (Wittkampf et al., 2011). Muñoz-Navarro et al. (2016) tested it in Spanish primary care settings and modified the original algorithm to increase the sensitivity for PD diagnosis: the most optimal cut-off point for screening purposes was 5 (the first item [for panic screening] and one of the following three, plus four somatic symptoms) (sensitivity of 77% and specificity of 72%).
Change in somatoform symptoms: 15-item Patient Health Questionnaire (PHQ-15) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The PHQ-15 (Kroenke et al., 2002) is the somatization module of the PHQ. It includes 13 somatic symptoms plus 2 from the PHQ-9 (sleeping problems and fatigue). Scores of 5, 10, and 15 represent low, medium, and high somatic symptom severity, respectively. To screen a somatization disorder, whereas the original algorithm needs of at least a score of 2 in three or more somatic symptoms (sensitivity of 78% and specificity of 71%) (van Ravesteijn et al., 2009), the cut point usually used is 10; nevertheless, since this can be obtained with ten symptoms of mild severity, we decided to join both criteria to screen the disorder. Furthermore, an absence of biological cause is also often required (since PHQ-15 does not distinguish between medically explained and unexplained symptoms) (Kroenke et al., 2002), but the self-administered nature of the PHQ-15 makes difficult to determine this. The PHQ-15 has been validated with Spanish psychiatric outpatients (α = .78) (Ros et al., 2010).

SECONDARY OUTCOMES:
Change in the level of impairment: Sheehan Disability Scale (SDS) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The SDS (Sheehan et al., 1996) is a self-administered test that measures the subjective symptom-related impairment with five 11-point Likert items. The three first items rate key areas in the past month: work, social life/leisure activities, and family life/home responsibilities. It has two additional items to assess stress level and perceived social support in the past week. We will use the Spanish version developed by Bobes et al. (1999), that has shown good properties with primary care population (α = .83) (Luciano et al., 2010). One, four, and seven are the cut points for mild, moderate, and high disability, respectively. A total score of 25 or more indicates a general high disability, and the patient will be asked by a clinical psychologist to confirm: 'Are you on sick leave?', 'Can you do the housework?', and 'Can you engage socially?' (one question per area).
Change in general quality of life: World Health Organization Quality of Life Instrument-Brief version (WHOQOL-BREF) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  Psychological, physical, social, and environmental domains will be assessed through the twenty-six 5-point Likert items of the WHOQOL-BREF (The WHOQOL Group, 1998b), the abbreviated version of the 100-item WHOQOL (WHOQOL-100) (The WHOQOL Group, 1998a). The more the participant scores, the better quality of life they have. The WHOQOL has been validated with Spanish population (Lucas-Carrasco, 2012; Rocha et al., 2012) and has shown good psychometric properties: α > .7 in psychological, physical, and environmental domains, though social domain's internal consistency varies from .58 (Rocha et al., 2012) to .75 (Lucas-Carrasco, 2012).
Change in ruminative responses: Ruminative Responses Scale (RRS) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The RRS (Nolen-Hoeksema & Morrow, 1991) was originally developed to measure the ruminative responses to depressed mood. It has been validated with Spanish population (Hervás, 2008), however, only the 5-item 'brooding' factor subscale (RRS-B) will be used in this trial (α = .79) (Muñoz-Navarro et al., 2021). The RRS-B scores from 1 ("almost never") to 4 ("almost always") how often the participant thinks as it is described in each item when they are discouraged, sad or depressed.
Change in worry: Penn State Worry Questionnaire (PSWQ) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The PSWQ (Meyer et al., 1990) measures the pathological worry as an uncontrollable and general state (i.e., as a GAD feature). It has been validated in Spain (Sandín et al., 2009) and, in this study, it will be used an 8-item abbreviated version (PSWQ-A) (Crittendon & Hopko, 2006) that has already showed good properties in primary care (α = .9) (Muñoz-Navarro et al., 2021). The PSWQ-A items rate how much worries affect the person from 1 ("not at all typical of me") to 5 ("very typical of me").
Change in attentional and interpretational biases: Inventory of Cognitive Activity in Anxiety Disorders (IACTA) and Questionnaire of Cognitive Distortions in Emotional Disorders (CDTE) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The IACTA was originally developed by Cano-Vindel (2001). It includes subscales that assess distortions according to Eysenck's four-factor theory (Eysenck, 2000). The abbreviated panic version (IACTA-PB; α = .87) (Muñoz-Navarro et al., 2021) will be used to measure attentional biases. It specifically scores from 0 ("almost never") to 4 ("almost always") how often the participant has certain cognitive distortions.
  The Questionnaire of Cognitive Distortions in Emotional Disorders (CDTE) (The PsicAP Group, unpublished) scores from 0 ("almost never") to 4 ("almost always") the frequency of certain cognitive biases in the main EDs (MDD, GAD, PD, and somatization disorder). It includes 16 items that measure the presence of four factors: sustained attention bias (α = .96), divided attention bias (α = .95), magnification interpretational bias (α = .94), and catastrophization interpretational bias (α = .96), with high levels of discriminant validity among the four EDs (ROC values > .8).
Change in emotion regulation strategies: Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The CERQ-36 (Garnefski et al., 2001) was developed for measuring the specific cognitive emotion regulation strategies that a person uses to face a stressful event. It scores from 1 ("almost never") to 5 ("almost always") how often the participant thinks as described. The CERQ has been validated with Spanish population (Domínguez-Sánchez et al., 2013) and the 27-item shortened version (Holgado-Tello et al., 2018) will be used (α values range from .72 ['acceptance'] to .88 ['positive refocus']).
Change in metacognitions: 30-item Metacognitions Questionnaire (MCQ-30) | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The MCQ-30 (Wells & Cartwright-Hatton, 2004) is a short form of the original MCQ (Cartwright-Hatton & Wells, 1997), which measures the beliefs about the own thinking processes. It has been validated with Spanish population (Ramos-Cejudo et al., 2013) and, in the current trial, only the 6-item 'negative beliefs' (about uncontrollability/danger) subscale (MCQ-NB; α = .82) will be used (Muñoz-Navarro et al., 2021). It scores from 1 ("totally disagree") to 4 ("totally agree") how the patient agrees with the sentences written.
Sociodemographic and medical data, and treatment satisfaction | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  An ad hoc questionnaire will be used to collect sociodemographic (gender, age, civil status, educative level, employment situation, and income level) and ED-related medical data (public and private health care consultations, accidents, medical tests, and sick leaves in the past 3 months; psychotropic drugs or other medication, and their posology), and it includes an additional question about treatment satisfaction (only at post-treatment and follow-ups). Medical records will be also consulted to complete the information (for privacy reasons, only strictly necessary data will be collected).
Cost and utility data | Baseline, immediately after the intervention, and follow-ups (6 and 12 months)
  The medical data collected will be used for cost calculations too. In addition, cost-utility will be measured through the European Quality of Life Scale (EuroQoL, EQ) (The EuroQol Group, 1990). The Spanish version of the 5-domain, 5-level EuroQol (EQ-5D-5L) (Badia et al., 1999; van Reenen et al., 2019) will be used to calculate the quality-adjusted life years (QALYs). The EQ-5D-5L measures five domains of health-related quality of life (mobility, self-care, daily activities, pain/unease, and anxiety/depression) through 5 severity levels ("no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems"), being able to stablish up to 3125 different health states, each of which can be represented through an index value that reflects the health state quality contextualized in the person's country/region. It also includes a visual analogue scale (VAS) that scores from 0 to 100 the current subjective, general health state.
Presence of eating disorders or alcohol abuse (exclusion criterion) | Pre-intervention (screening)
  The PHQ also lets to measure the presence of other mental disorders. The Spanish version (Díez-Quevedo et al., 2001) detects eating disorders, such as bulimia nervosa or binge eating disorder, with a sensitivity of 92% and a specificity of 98%; and alcohol abuse with a sensitivity of 76% and a specificity of 99%. Affirmative answers to items 6a to 6c and 8 indicate bulimia nervosa; if item 8 were answered negatively (or unanswered), it would point out a binge eating disorder. An affirmative answer to any of the items 10a to 10e would indicate alcohol abuse. In any of these cases the patient would be interviewed by a clinical psychologist to confirm a possible diagnosis of eating, alcohol or personality disorder.

OTHER OUTCOMES:
Presence of emotional disorder (inclusion criterion): Patient Health Questionnaire 4 items (PHQ-4) | Pre-intervention (screening)
  The PHQ-4 (Kroenke et al., 2009) will be used for the recruitment phase. The PHQ-4 gathers the two items from the PHQ-2 and the two from the GAD-2 (short versions of the PHQ-9 and GAD-7, respectively). It has been studied with Spanish primary care population (Spearman-Brown's ρ[PHQ-4] = .72; ρ[PHQ-2] = .86; ρ[GAD-2] = .76) (Cano-Vindel et al., 2018): a score greater than or equal to 3 would indicate a need of additional assessment (PHQ-2: sensitivity of 90%, specificity of 61%; GAD-2: sensitivity of 88%, specificity of 61%). It may be an extremely useful tool, as it helps to accelerate the screening process, however, it has been suggested that both PHQ-2 and GAD-2 sum scores should be regarded separately in primary care samples (Cano-Vindel et al., 2018). The first item from the PHQ-PD has been added to screen panic disorder.
Presence of severe mental disorders (exclusion criterion) | Pre-intervention (screening)
  In the case of scoring as a severe ED (depressive or anxiety disorder) or other mental illness in the PHQ, or when the diagnosis is not clear, the patient will undergo a second evaluation with a gold-standard tool. The Structured Clinical Interview for DSM Axis-I Disorders (SCID-I) (First et al., 1999) will be used to assess panic and depression disorders, whereas the Composite International Diagnostic Interview (CIDI) (WHO's Mental Health Division, 1997) will be used for GAD (since the former may not be adequate as it only includes one item for GAD).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Moriana Elvira, PhD, Principal Investigator — Universidad de Córdoba
Locations (3):
- Spain (3):
  - Unidad de Salud Mental Comunitaria Montilla, Montilla, Córdoba
  - Centro Sanitario "Levante Sur Dr. Manuel Barragán Solís", Córdoba
  - Centro Sanitario "Carlos Castilla del Pino", Córdoba

REFERENCES:
- [Background] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Background] Barlow DH, Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Allen LB, et al. Protocolo Unificado para el Tratamiento Transdiagnóstico de los Trastornos Emocionales [Unified Protocol for Transdiagnostic Treatment of Emotional Disorders: Therapist Guide and Patient Guide]. 1st ed. Alianza; 2015.
- [Background] Bobes J, Badia X, Luque A, Garcia M, Gonzalez MP, Dal-Re R. [Validation of the Spanish version of the Liebowitz social anxiety scale, social anxiety and distress scale and Sheehan disability inventory for the evaluation of social phobia]. Med Clin (Barc). 1999 Apr 24;112(14):530-8. Spanish. PMID 10363239
- [Background] Cano-Vindel A. [Inventory of Cognitive Activity in Anxiety Disorders (IACTA)]. Unpublished; 2001.
- [Background] Cano-Vindel A, Munoz-Navarro R, Medrano LA, Ruiz-Rodriguez P, Gonzalez-Blanch C, Gomez-Castillo MD, Capafons A, Chacon F, Santolaya F; PsicAP Research Group. A computerized version of the Patient Health Questionnaire-4 as an ultra-brief screening tool to detect emotional disorders in primary care. J Affect Disord. 2018 Jul;234:247-255. doi: 10.1016/j.jad.2018.01.030. Epub 2018 Feb 16. PMID 29549826
- [Background] Cartwright-Hatton S, Wells A. Beliefs about worry and intrusions: the Meta-Cognitions Questionnaire and its correlates. J Anxiety Disord. 1997 May-Jun;11(3):279-96. doi: 10.1016/s0887-6185(97)00011-x. PMID 9220301
- [Background] Clark DM. Realizing the Mass Public Benefit of Evidence-Based Psychological Therapies: The IAPT Program. Annu Rev Clin Psychol. 2018 May 7;14:159-183. doi: 10.1146/annurev-clinpsy-050817-084833. Epub 2018 Jan 19. PMID 29350997
- [Background] Crittendon J, Hopko DR. Assessing worry in older and younger adults: Psychometric properties of an abbreviated Penn State Worry Questionnaire (PSWQ-A). J Anxiety Disord. 2006;20(8):1036-54. doi: 10.1016/j.janxdis.2005.11.006. Epub 2006 Jan 4. PMID 16387472
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Dominguez-Sanchez FJ, Lasa-Aristu A, Amor PJ, Holgado-Tello FP. Psychometric properties of the Spanish version of the Cognitive Emotion Regulation Questionnaire. Assessment. 2013 Apr;20(2):253-61. doi: 10.1177/1073191110397274. Epub 2011 Apr 5. PMID 21467092
- [Background] Eysenck MW. A cognitive approach to trait anxiety. Eur J Pers. 2000 Sep;14(5):463-76
- [Background] First MB, Spitzer RL, Gibbon M, Williams JBW. Entrevista Clínica Estructurada para los Trastornos del Eje I del DSM-IV. Barcelona: Masson; 1999.
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Garnefski N, Kraaij V, Spinhoven P. Negative life events, cognitive emotion regulation and emotional problems. Pers Individ Dif. 2001;30(8):1311-27.
- [Background] González-Blanch C, Umaran-Alfageme O, Cordero-Andrés P, Muñoz-Navarro R, Ruiz-Rodríguez P, Medrano LA, et al. Tratamiento psicológico de los trastornos emocionales en Atención Primaria: el manual de tratamiento transdiagnóstico del estudio PsicAP. Ansiedad y Estrés. 2018;24(1).
- [Background] Hervás G. Adaptación al castellano de un instrumento para evaluar el estilo rumiativo: la Escala de Respuestas Rumiativas. Rev Psicopatología y Psicol Clínica. 2008;13(2):111-21.
- [Background] Holgado-Tello FP, Amor PJ, Lasa-Aristu A, Domínguez-Sánchez FJ, Delgado B. Two new brief versions of the Cognitive Emotion Regulation Questionnaire and its relationships with depression and anxiety. An Psicol. 2018;34(3):458-64.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Lucas-Carrasco R. The WHO quality of life (WHOQOL) questionnaire: Spanish development and validation studies. Qual Life Res. 2012 Feb;21(1):161-5. doi: 10.1007/s11136-011-9926-3. Epub 2011 May 25. PMID 21611868
- [Background] Luciano JV, Bertsch J, Salvador-Carulla L, Tomas JM, Fernandez A, Pinto-Meza A, Haro JM, Palao DJ, Serrano-Blanco A. Factor structure, internal consistency and construct validity of the Sheehan Disability Scale in a Spanish primary care sample. J Eval Clin Pract. 2010 Oct;16(5):895-901. doi: 10.1111/j.1365-2753.2009.01211.x. PMID 20626541
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Muñoz-Navarro R, Adrián Medrano L, González-Blanch C, Carpallo-González M, Olave L, Iruarrizaga I, et al. Validity of Brief Scales for Assessing Transdiagnostic Cognitive Emotion Regulation Strategies in Primary Care Patients With Emotional Disorders. Eur J Psychol Assess. 2021;37(2):86-94.
- [Background] Munoz-Navarro R, Cano-Vindel A, Medrano LA, Schmitz F, Ruiz-Rodriguez P, Abellan-Maeso C, Font-Payeras MA, Hermosilla-Pasamar AM. Utility of the PHQ-9 to identify major depressive disorder in adult patients in Spanish primary care centres. BMC Psychiatry. 2017 Aug 9;17(1):291. doi: 10.1186/s12888-017-1450-8. PMID 28793892
- [Background] Munoz-Navarro R, Cano-Vindel A, Moriana JA, Medrano LA, Ruiz-Rodriguez P, Aguero-Gento L, Rodriguez-Enriquez M, Piza MR, Ramirez-Manent JI. Screening for generalized anxiety disorder in Spanish primary care centers with the GAD-7. Psychiatry Res. 2017 Oct;256:312-317. doi: 10.1016/j.psychres.2017.06.023. Epub 2017 Jun 12. PMID 28666201
- [Background] Munoz-Navarro R, Cano-Vindel A, Wood CM, Ruiz-Rodriguez P, Medrano LA, Limonero JT, Tomas-Tomas P, Gracia-Gracia I, Dongil-Collado E, Iruarrizaga MI; PsicAP Research Group. The PHQ-PD as a Screening Tool for Panic Disorder in the Primary Care Setting in Spain. PLoS One. 2016 Aug 15;11(8):e0161145. doi: 10.1371/journal.pone.0161145. eCollection 2016. PMID 27525977
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Ramos-Cejudo J, Salguero JM, Cano-Vindel A. Spanish version of the Meta-Cognitions Questionnaire 30 (MCQ-30). Span J Psychol. 2013;16:E95. doi: 10.1017/sjp.2013.95. PMID 24230958
- [Background] Rocha NS, Power MJ, Bushnell DM, Fleck MP. Cross-cultural evaluation of the WHOQOL-BREF domains in primary care depressed patients using Rasch analysis. Med Decis Making. 2012 Jan-Feb;32(1):41-55. doi: 10.1177/0272989X11415112. Epub 2011 Aug 8. PMID 21825270
- [Background] Ros Montalban S, Comas Vives A, Garcia-Garcia M. Validation of the Spanish version of the PHQ-15 questionnaire for the evaluation of physical symptoms in patients with depression and/or anxiety disorders: DEPRE-SOMA study. Actas Esp Psiquiatr. 2010 Nov-Dec;38(6):345-57. Epub 2010 Nov 1. PMID 21188674
- [Background] Sandín B, Chorot P, Valiente RM, Lostao L. Validación española del cuestionario de preocupación PSWQ: estructura factorial y propiedades psicométricas. Rev Psicopatología y Psicol Clínica. 2009;14(2):107-22.
- [Background] Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996 Jun;11 Suppl 3:89-95. doi: 10.1097/00004850-199606003-00015. PMID 8923116
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] The PsicAP Group. Cuestionario de Distorsiones Cognitivas en Trastornos Emocionales (CDTE) [Questionnaire of Cognitive Distortions in Emotional Disorders (CDTE)]. Unpublished;
- [Background] The World Health Organization Quality of Life Assessment (WHOQOL): development and general psychometric properties. Soc Sci Med. 1998 Jun;46(12):1569-85. doi: 10.1016/s0277-9536(98)00009-4. PMID 9672396
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] van Ravesteijn H, Wittkampf K, Lucassen P, van de Lisdonk E, van den Hoogen H, van Weert H, Huijser J, Schene A, van Weel C, Speckens A. Detecting somatoform disorders in primary care with the PHQ-15. Ann Fam Med. 2009 May-Jun;7(3):232-8. doi: 10.1370/afm.985. PMID 19433840
- [Background] van Reenen M, Janssen B, Stolk E, Secnik Boye K, Herdman M, Kennedy-Martin M, et al. EQ-5D-5L User Guide. 3.0. EuroQol Research Foundation; 2019. Available from: https://euroqol.org/publications/user-guides/
- [Background] Watts SE, Turnell A, Kladnitski N, Newby JM, Andrews G. Treatment-as-usual (TAU) is anything but usual: a meta-analysis of CBT versus TAU for anxiety and depression. J Affect Disord. 2015 Apr 1;175:152-67. doi: 10.1016/j.jad.2014.12.025. Epub 2014 Dec 15. PMID 25618002
- [Background] Wells A, Cartwright-Hatton S. A short form of the metacognitions questionnaire: properties of the MCQ-30. Behav Res Ther. 2004 Apr;42(4):385-96. doi: 10.1016/S0005-7967(03)00147-5. PMID 14998733
- [Background] WHO's Mental Health Division. Entrevista Diagnóstica Internacional Compuesta (CIDI). Geneva, Switzerland: World Health Organization; 1997.
- [Background] Wittkampf KA, Baas KD, van Weert HC, Lucassen P, Schene AH. The psychometric properties of the panic disorder module of the Patient Health Questionnaire (PHQ-PD) in high-risk groups in primary care. J Affect Disord. 2011 Apr;130(1-2):260-7. doi: 10.1016/j.jad.2010.10.030. Epub 2010 Nov 13. PMID 21075451
- [Derived] Aguilera-Martin A, Galvez-Lara M, Cuadrado F, Moreno E, Garcia-Torres F, Vencesla JF, Corpas J, Jurado-Gonzalez FJ, Munoz-Navarro R, Gonzalez-Blanch C, Ruiz-Rodriguez P, Barrio-Martinez S, Prieto-Vila M, Carpallo-Gonzalez M, Cano-Vindel A, Moriana JA. Cost-effectiveness and cost-utility evaluation of individual vs. group transdiagnostic psychological treatment for emotional disorders in primary care (PsicAP-Costs): a multicentre randomized controlled trial protocol. BMC Psychiatry. 2022 Feb 9;22(1):99. doi: 10.1186/s12888-022-03726-4. PMID 35139809